CLINICAL TRIAL: NCT06928870
Title: The Effect of Controlled Hypotension on Cerebral Oxygen Saturation in Spinal Surgery
Brief Title: The Effect of Controlled Hypotension
Acronym: NIRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Damla Usalan, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AEŞH-EK1-2024-0003
Record Dates: First submitted 2025-02-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Hypoperfusion; Hypotension
Keywords: cerebral oxygen saturation; NIRS; controlled hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group MAP 55-65 mmHg (Other): Group - MAP 55-65 mmHg: MAP will be maintained between 55-65 mmHg during anesthesia.
  Interventions: Other: MAP 55-65 mmHg
- Group MAP 66-75 mmHg (Other): Group - MAP 66-75 mmHg: MAP will be maintained between 66-75 mmHg during anesthesia.
  Interventions: Other: MAP 66-75 mmHg

INTERVENTIONS:
Other: MAP 55-65 mmHg — MAP will be maintained between 55-65 mmHg during anesthesia.
  Arms: Group MAP 55-65 mmHg
Other: MAP 66-75 mmHg — MAP will be maintained between 66-75 mmHg during anesthesia.
  Arms: Group MAP 66-75 mmHg

SUMMARY:
Controlled hypotension is currently used in spinal surgery to reduce bleeding at the surgical site, improve the surgeon's visibility, and decrease intraoperative blood loss. Although controlled hypotension is considered a beneficial method from a surgical perspective, it is important to be cautious about its side effects. One such side effect is cerebral perfusion insufficiency, which can be managed by monitoring cerebral circulation through regional cerebral oxygen saturation (rSO2).

The aim of this study is to compare the effects of controlled hypotension at specific MAP ranges on cerebral oxygen saturation.

DETAILED DESCRIPTION:
Controlled hypotension is currently used in spinal surgery to reduce bleeding at the surgical site, improve the surgeon's visibility, and decrease intraoperative blood loss. Although controlled hypotension is considered a beneficial method from a surgical perspective, it is important to be cautious about its side effects. One such side effect is cerebral perfusion insufficiency, which can be managed by monitoring cerebral circulation through regional cerebral oxygen saturation (rSO2).

In the literature, various definitions of controlled hypotension exist. It is commonly defined as maintaining the Mean Arterial Pressure (MAP) between 50-65 mmHg, Systolic Arterial Pressure (SAP) between 80-90 mmHg, or reducing MAP by 30% compared to baseline values. In our study, we plan to maintain the MAP within the range of 55-75 mmHg and compare the effects of two different MAP levels on perioperative cerebral oxygen saturation, anesthetic and surgical parameters, and postoperative cognitive functions.

The aim of this study is to compare the effects of controlled hypotension at specific MAP ranges on cerebral oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* ASA I-III risk group
* BMI between 18-40
* Baseline blood pressure below 140/90 mmHg
* Scheduled to undergo spinal surgery (2-4 level instrumentation)

Exclusion Criteria:

* Below 18 or above 65 years old
* Advanced comorbidities
* ASA IV or higher
* Baseline blood pressure above 140/90 mmHg
* History of bleeding diathesis
* Use of anticoagulant medications
* BMI below 18 or above 40
* History of previous spinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Near infrared spectroscopy (NIRS) | 5 minutes before induction of anesthesia
  cerebral oxygen saturation
Near infrared spectroscopy (NIRS) | 5 minutes after intubation
  cerebral oxygen saturation
Near infrared spectroscopy (NIRS) | 5 minutes after positioning prone
  cerebral oxygen saturation
Near infrared spectroscopy (NIRS) | 1 minutes after first surgical incision is made
  cerebral oxygen saturation
Near infrared spectroscopy (NIRS) | the time after one minutes target MAP value
  cerebral oxygen saturation
Near infrared spectroscopy (NIRS) | the time after ten minutes target MAP value
  cerebral oxygen saturation
Near infrared spectroscopy (NIRS) | the time after 20 minutes target MAP value
  cerebral oxygen saturation
Near infrared spectroscopy (NIRS) | 5 minutes after extubation
  cerebral oxygen saturation
Near infrared spectroscopy (NIRS) | postextubation after 15 minutes
  cerebral oxygen saturation

SECONDARY OUTCOMES:
mini mental test | 15 minutes before induction of anesthesia
  It is used to evaluate cognitive function.
mini mental test | 30 minutes after extubation
  It is used to evaluate cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: damla usalan, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Varlık Mahallesi Yenimahalle, Turkey (Türkiye)

REFERENCES:
- [Background] Dutton RP. Controlled hypotension for spinal surgery. Eur Spine J. 2004 Oct;13 Suppl 1(Suppl 1):S66-71. doi: 10.1007/s00586-004-0756-7. Epub 2004 Jun 9. PMID 15197633
- [Result] Ooms M, Schooss R, Winnand P, Heitzer M, Holzle F, Bickenbach J, Rieg A, Modabber A. Influence of perioperative blood pressure regulation on postoperative delirium in patients undergoing head and neck free flap reconstruction. Eur J Med Res. 2023 Sep 22;28(1):365. doi: 10.1186/s40001-023-01367-1. PMID 37736691